CLINICAL TRIAL: NCT04899310
Title: A Global Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of mRNA-3705 in Participants With Isolated Methylmalonic Acidemia Due to Methylmalonyl-CoA Mutase Deficiency
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of mRNA-3705 in Participants With Isolated Methylmalonic Acidemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mRNA-3705-P101; 2022-502492-32-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Methylmalonic Acidemia
Keywords: Isolated Methylmalonic Acidemia; Isolated Methylmalonic Aciduria; Elevated Methylmalonic Acid (MMA); Metabolism, Inborn Errors; Genetic Diseases; Moderna; mRNA; mRNA-3705
MeSH Terms: conditions — Methylmalonic acidemia; Metabolism, Inborn Errors; Genetic Diseases, Inborn | interventions — Methylmalonyl-CoA Mutase

STUDY DESIGN:
Intervention Model Description: Parts 2 and 3 run in parallel and occur after Part 1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Parts 1 and 3 are open label and non-randomized. Part 2 is blinded and randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- mRNA-3705 (Experimental): Participants in Part 1 will receive a weight-based dose of mRNA-3705, administered IV, once every 2 weeks or once every 3 weeks for up to 10 doses over approximately 40 weeks. Participants in Part 2 and Part 3 will receive mRNA-3705 at the selected dose level and frequency for 3 months.
  Interventions: Biological: mRNA-3705
- Placebo (Placebo Comparator): Participants only in Part 2 will receive placebo at the selected frequency for 3 months.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-3705 — Sterile liquid for infusion
  Other Names: modified mRNA encoding human; methylmalonyl-coenzyme A mutase
  Arms: mRNA-3705
Biological: Placebo — Sterile liquid for infusion
  Arms: Placebo

SUMMARY:
This is a study of mRNA-3705 in participants with isolated elevated methylmalonic acid (MMA) due to methylmalonyl-coenzyme A (CoA) mutase (MUT) deficiency. The main goal of the study is to assess safety, efficacy, pharmacokinetics, and pharmacodynamics of intravenously (IV)-infused mRNA-3705.

DETAILED DESCRIPTION:
This study comprises 3 parts and is designed to evaluate multiple doses and dosing intervals of mRNA-3705.

Parts 1 and 3 are designed to characterize the safety, tolerability, and pharmacological activity of mRNA-3705 administered via intravenous infusion to participants with isolated MMA due to MUT deficiency. Part 2 will evaluate the efficacy of mRNA-3705 as assessed by the change in plasma methylmalonic acid levels.

Participants who complete the treatment period in any part of the study, including the end of treatment (EOT) visit, will be offered participation in the mRNA-extension study (mRNA-3705-P101-EXT; NCT05295433) or may transition to the follow-up period of the study. All participants, including those randomized to placebo in Part 2, will receive mRNA-3705 in the extension study.

ELIGIBILITY:
Key Inclusion Criteria:

* (Part 1 only) Participant has a body weight of ≥11.0 kilograms at the screening visit.
* Participant has a diagnosis of isolated MMA due to MUT deﬁciency conﬁrmed by molecular genetic testing.
* Participant has a blood vitamin B12 level equal to or above the lower limit of normal (based on laboratory reference range) conﬁrmed in the screening period.
* Participant or their legally authorized representative is willing and able to provide informed consent and/or assent as mandated by local regulations and is willing and able to comply with study-related assessments.
* Sexually active participants of childbearing or reproductive potential agree to use a highly effective method of contraception, consistent with local regulations, during the study and for 3 months after the last administration of study drug.
* (Part 2 only) Participants with 2 screening MMA levels ≥400 micromolar.
* (Parts 2 and 3 only) Participant is ≥5 years of age at the time of informed consent/assent.

Key Exclusion Criteria:

* Participant has a diagnosis of isolated MMA cofactor adenosyl-cobalamin (cb1A, cb1B, or cb1D) enzymatic subtypes or methylmalonyl-CoA epimerase deficiency or combined MMA with homocystinuria.
* Participant has previously received gene therapy for the treatment of MMA.
* Participant has a history of organ transplantation or planned organ transplantation during the period of study participation.
* Participant has an active, unstable, or clinically significant medical condition not related to MMA or history of noncompliance that, in the investigator's opinion, could potentiate the risk while participating in this study, interfere with the interpretation of study results, or limit the participant's participation in the study. This may include, but is not limited to, history of relevant food or drug allergies; history of cardiovascular, central nervous, gastrointestinal, or infectious disease; history of clinically significant pathology; and/or history of cancer.
* (Part 2 only) Participant has the partial MUT deficiency disease phenotype, as assessed by genotyping, clinical phenotype/presentation, or vitamin B12-responsive MMA.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 3: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Study Drug-related TEAEs, Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), and TEAEs Leading to Treatment Discontinuation | Up to 134 weeks
Part 2: Percentage Change in Plasma MMA Levels at Month 3 | Baseline, Month 3

SECONDARY OUTCOMES:
Parts 1 and 3: Percentage Change in Plasma MMA Level | Baseline up to Week 30
Part 1: Maximum Observed Effect (Emax) for Plasma MMA Measurement after Single and Repeated Administrations of mRNA-3705 | Baseline up to Week 30
Part 1: Area Below the Baseline and Above the Response Curve (AUC_Below_B) for Plasma MMA Measurement after Single and Repeated Administrations of mRNA-3705 | Baseline up to Week 30
Part 1: Area Under the Curve that is the Area Under the Response Curve Above the Baseline (AUC_Above_B)-AUC_Below_B (AUC_Net_B) for Plasma MMA Measurement after Single and Repeated Administrations of mRNA-3705 | Baseline up to Week 30
Parts 1-3: Percentage Change in Plasma 2-Methylcitric Acid (2-MC) Levels | Baseline up to Week 30
Parts 1-3: Maximum Observed Concentration (Cmax) of human Methylmalonyl-Coenzyme A Mutase (hMUT) mRNA-3705 | 0 (predose) to 264 hours postdose
Parts 1-3: Area Under the Concentration-Time Curve (AUC) of hMUT mRNA-3705 | 0 (predose) to 264 hours postdose
Parts 1-3: Titer of Anti-Polyethylene Glycol (PEG) Antibodies | 0 (predose) to 336 hours postdose
Parts 2 and 3: Titer of Anti-hMUT Antibodies | 0 (predose) to 336 hours postdose
Parts 2 and 3: Change from Baseline in Pediatric Quality of Life Inventory (PedsQL) Physical Function Score | Baseline, Month 3
Parts 2 and 3: Annualized Frequency of MMA-related Hospitalizations | Baseline up to Month 3
Parts 2 and 3: Annualized Frequency of Metabolic Decompensation Events | Baseline up to Month 3
Parts 2 and 3: Change from Baseline in PedsQL Total Score | Baseline, Week 47
Parts 2 and 3: Change from Baseline in Investigator Global Assessment of Severity (IGA-S) | Baseline, Week 47
Parts 2 and 3: Change from Baseline in Caregiver-Reported Global Impression of Severity (CrGI-S) | Baseline, Week 47
Parts 2 and 3: Change from Baseline in Investigator Global Assessment of Improvement (IGA-I) | Week 3 (Dose 2), Week 47
Parts 2 and 3: Change from Baseline in Caregiver-Reported Global Impression of Improvement (CrGI-I) | Week 3 (Dose 2), Week 47
Part 2: Number of Participants with TEAEs, SAEs, AESIs, and TEAEs Leading to Treatment Discontinuation | Up to 47 weeks
Part 2: Plasma Concentration of SM-86 | 0 (predose) to 48 hours postdose

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Canada (2):
  - Stollery Children's Hospital University of Alberta, Edmonton, Alberta
  - Hospital For Sick Children, Toronto, Ontario
- Hôpital Necker - Enfants Malades, Paris, France
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (2):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitario 12 de Octubre, Madrid
- Royal Manchester Children's Hospital, Manchester, United Kingdom